CLINICAL TRIAL: NCT06356298
Title: Airway Management Effects of Flexible Reinforced Laryngeal Mask Airway Versus Endotracheal Tube for Childhood Adenotonsillectomy：a Randomized Controlled Trial
Brief Title: Flexible Reinforced Laryngeal Mask Airway Versus Endotracheal Tube for Childhood Adenotonsillectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy Chief Physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MCHH_004
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia Intubation Complication; Airway; Adenotonsillectomy; Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLMA group (Experimental): In the FLMA group, a FLMA was applied.
  Interventions: Other: Airway Management: Flexible Reinforced Laryngeal Mask Airway
- ETT group (Experimental): In the ETT group, guided by a visual laryngoscope, a ETT was intubated.
  Interventions: Other: Airway Management: Endotracheal Tube

INTERVENTIONS:
Other: Airway Management: Flexible Reinforced Laryngeal Mask Airway — In the FLMA group, a FLMA was applied according to the manufacturer's recommendations. After lubrication of the posterior surface with oxybuprocaine hydrochloride gel, the FLMA was inserted after propping the shoulders. Its cuff was fully deflated before insertion, and the pressure was adjusted to 40 cm H2O with a manometer after insertion.
  Arms: FLMA group
Other: Airway Management: Endotracheal Tube — In the ETT group, guided by a visual laryngoscope, a ETT was intubated after lubrication of the surface with oxybuprocaine hydrochloride gel: endotracheal tube size = (16+ age) /4. The cuff pressure of ETT was adjusted to 20 cm H2O with a handheld manometer after inflation.
  Arms: ETT group

SUMMARY:
The goal of this clinical trial is to compare the airway management effects of flexible reinforced laryngeal mask and endotracheal tube in childhood adenotonsillectomy.

Participants will be randomly allocated to two groups: endotracheal tube group (ETT) and flexible reinforced laryngeal mask group (FLMA). For those in ETT group: they will be intubated after induction of anesthesia .For those in FLMA group: they will be put in flexible reinforced laryngeal mask after induction of anesthesia .

The investigators will compare FLMA with ETT to see if flexible reinforced laryngeal mask can be used safely and effectively in childhood adenotonsillectomy，and if there will be less severe adverse events in FLMA.

ELIGIBILITY:
Inclusion Criteria:

* patients who choose to have adenotonsillectomy surgery
* the American Society of Anesthesiologists (ASA) physical status ranked I-II
* the oropharyngeal anatomy is normal
* competent to provide informed consent

Exclusion Criteria:

* upper respiratory tract infection one week before surgery
* oropharyngeal anatomy is abnormal
* high risk of reflux aspiration
* liver or kidney failure
* psychiatric disorders

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Peak airway pressure | intraoperative period,10 minutes-1 hours
  Maximum peak airway pressure during surgery
Petco2 | intraoperative period,10 minutes-1 hour
  Petco2 at the end of surgery
Ventilation leakage or not | intraoperative period,10 minutes-1 hour
  Using volume ventilation, tidal volume set to 10 ml /kg, Ventilation leakage is defined as reaching more than 20% of the set tidal volume.

SECONDARY OUTCOMES:
Mean arterial pressure (MAP) | Intraoperative period, 30 minutes - 1.5 hours
  MAP level will be monitored and recorded at 6 time points, including the entry into the operation room (Time 0), 2 min after anesthesia induction (Time 1), implantation of FLMA or ETT (Time 2), implantation of mouth opener (Time 3) ，at the end of surgery (Time 4), and after removal of FLMA or ETT (Time 5)
Heart rate (HR) | Intraoperative period, 30 min - 1.5 hours
  HR will be monitored and recorded at 4 time points, including the entry into the operation room (Time 0), 2 min after anesthesia induction (Time 1), implantation of FLMA or ETT (Time 2), implantation of mouth opener (Time 3) ，at the end of surgery (Time 4), and after removal of FLMA or ETT (Time 5)
Recovery time | Postoperative 30 minutes
  Time to fully awake, defined as by a modified Aldrete score which will be recorded every 3 minutes from the end of the procedure with a recovery index (MAS) of 9 or more.
Extubation time | Postoperative 30 minutes
  Time to extubate, defined as occurrence of regular respiration from the end of the procedure.
Dosage of anesthetic | Intraoperative period, 30 minutes - 1.5 hours
  The total amount of sedative and analgesic drugs will be recorded.
Success of FLMA or ETT | Intraoperative period, 10 minutes - 1hour
  The first success of FLMA or ETT rate will be recorded, and insertion over three times will be considered as failed intubation.
Surgeon satisfaction | Postoperative 30 minutes
  Record the satisfaction of the surgeon with the FLMA or ETT, defined as a score out of100.
Adverse events | Postoperative 1 hour
  The adverse events will be monitored and recorded during the operation and post-operation. AE will include: nausea and vomiting, reflux aspiration, hoarseness, dysphagia, sore throat, coughing, bronchospasm, laryngeal spasm, mask with blood, respiratory depression (defined as SpO2< 90%),

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei, China